CLINICAL TRIAL: NCT01248078
Title: Antibiotic Prophylaxis Before Surgery Versus After Cord Clamping in Elective Cesarean Delivery - a Double-blind, Prospective, Randomized Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Armin Witt, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 226/2003
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Elective Cesarean Section
Keywords: elective cesarean section; antibiotic prophylaxis; cefazoline; wound infection
MeSH Terms: conditions — Wound Infection | interventions — Cephalexin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cefazolin A (Active Comparator): administered before skin incision
  Interventions: Drug: Keflex
- Cefazolin B (Active Comparator): after umbilical cord clamping
  Interventions: Drug: Keflex
- saline solution (Placebo Comparator): administered before skin incision
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Keflex — 2g of i.v. cefazolin singleshot administered before skin incision
  Arms: Cefazolin A
Drug: Keflex — 2g of i.v. cefazolin singleshot administered after umbilical cord clamping
  Arms: Cefazolin B
Drug: saline solution — 100cc administered before skin incision
  Arms: saline solution

SUMMARY:
In this prospective, randomized, placebo controlled trial the investigators were able to demonstrate the usefulness of prophylactic cefazolin in elective caesarean section versus placebo, irrespective of the timing of administration, ie before skin incision or after umbilical cord clamping

DETAILED DESCRIPTION:
Background. Perioperative antibiotic prophylaxis during elective cesarean section at term to reduce postoperative maternal infectious morbidity is generally used but may not be efficient based on the available data. Also, the optimal timing of prophylactic antibiotic administration is unclear.

Methods. The investigators compared the effectiveness of cefazolin, administered before skin incision versus after umbilical cord clamping versus placebo in a three-arm randomized trial. The primary endpoint of the study was postoperative infectious morbidity, defined as wound infection, endometritis, or urinary tract infection. Results: The primary outcome was observed in 18/370 women in group 1 (4.9%) and in 14/371 women in group 2 (3.8%), whereas it was noted in 45/371 women in group 3 (12.1%; p<0.001 for group 1 vs. group 3; p<0.001 for group 2 vs. group 3; p<0.001 for group 1 vs. group 2 vs. group 3). The number needed to treat to avoid one primary outcome was 13. Comparing groups 1 and 2, there was no statistically significant difference regarding the primary outcome (p=0.6).

Conclusions. In this prospective, randomized, placebo controlled trial the investigators were able to demonstrate the usefulness of prophylactic cefazolin in elective caesarean section versus placebo, irrespective of the timing of administration, ie before skin incision or after umbilical cord clamping.

ELIGIBILITY:
Inclusion Criteria:

- Elective cesarean section at term Patientin >18 years Informed consent NO known allergy to cefazolin NO exposure to any antibiotic agent within 1 week prior to delivery

Exclusion Criteria:

- cesarean section before week 37 cephalosporin allergy age less than 18 years exposure to any antibiotic agent within 1 week prior to delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1112 (Actual)
Dates: Start 2004-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
postoperative infectious morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Witt A, Doner M, Petricevic L, Berger A, Germann P, Heinze G, Tempfer C. Antibiotic prophylaxis before surgery vs after cord clamping in elective cesarean delivery: a double-blind, prospective, randomized, placebo-controlled trial. Arch Surg. 2011 Dec;146(12):1404-9. doi: 10.1001/archsurg.2011.725. PMID 22184305